CLINICAL TRIAL: NCT02038205
Title: High Resolution Ultrasonographic Measurements of the Median Nerve Before and After Wrist Splinting for Carpal Tunnel Syndrome
Brief Title: Ultrasonographic Measurements of the Median Nerve Before and After Splinting for Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 336315
Record Dates: First submitted 2014-01-07; First posted 2014-01-16 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
A prospective cohort follow-up study design is undertaken. Both males and females with mild to moderate carpal tunnel syndrome will receive standard-of-care wrist splint for 6 weeks and undergo follow up studies for data collection. Controls will also be seen for a one time visit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older and;
* Diagnosis of mild to moderate CTS with median motor latency at 8 cm is greater than 4.5 milliseconds or Combined Sensory Index > 0.9 where first line therapy is indicated to include nocturnal wrist bracing
* Control subjects without symptoms of carpal tunnel syndrome.

Exclusion Criteria:

* Evidence of severe CTS as seen with electromyographic changes in the body of the muscle
* Untreated hypothyroidism, Rheumatologic disorders
* Diagnosed Severe CTS or Chronic symptoms of carpal tunnel, greater than 1 year, this includes wasting of the hand muscles
* Undergoing or previously treated for carpal tunnel on affected side. This includes surgery (carpal tunnel release), corticosteroid injections, bracing within the last 3 months while wearing the brace consistently every night, or any other intervention.
* Currently pregnant or < 3 months post partum
* History of wrist, hand fracture or severe trauma to affected hand and/or wrist
* Known tumor, mass or deformity of the hand/wrist
* Inflammatory articular disease of the joints or tendons Existing cervical radiculopathy or previous surgeries to the neck for radicular symptoms
* History of electrodiagnostic evidence of generalized polyneuropathy or evidence of denervation
* Diagnosed neuromuscular disorders which may complicate CTS diagnosis
* Implanted electronic device (pacemaker, intrathecal pump/stimulator)
* Any illness that makes it unsafe for the patient to participate in the study
* Not fluent in English as NeuroQOL and other subjective information is limited to the English language interpretation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those with diagnosis of carpal tunnel syndrome, and healthy control subjects with no symptoms of CTS.
Sampling Method: Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Cross sectional area of median nerve using ultrasound | 6 weeks

SECONDARY OUTCOMES:
Patient-reported outcome measures using NeuroQOL and CTSAQ | 6 weeks
Motor latency, motor amplitude, sensory velocity and sensory amplitude with electrodiagnostic study | 6 weeks
cross sectional area, electrodiagnostic study, age, gender, height, weight, BMI, wrist circumference, wrist width. smoking and handedness as predictors of improvement (or no improvement) in the NeuroQOL and CTSAQ-measured clinical severity scale. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nanette Joyce, DO, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States